CLINICAL TRIAL: NCT03035188
Title: A Phase II, Single-armed, Multicenter Trial of Neoadjuvant Vismodegib in Patients With Large and/or Recurrent Resectable Basal Cell Carcinoma
Brief Title: Neoadjuvant Vismodegib in Patients With Large and/or Recurrent Resectable Basal Cell Carcinoma
Acronym: NICCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SRH Wald-Klinikum Gera GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADO-EP02 (ML29328)
Record Dates: First submitted 2016-12-26; First posted 2017-01-27 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2019-03

CONDITIONS: Basal Cell Carcinoma
Keywords: resectable
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vismodegib (Experimental): Continuous once-daily oral dosing of vismodegib at a dosage of 150 mg per administration
  Interventions: Drug: Vismodegib

INTERVENTIONS:
Drug: Vismodegib — 1 capsule (150 mg vismodegib) taken once daily for a maximum of 12 weeks.
  Other Names: Erivedge

SUMMARY:
In this study patients with resectable basal cell carcinoma (BCC) who usually undergo surgery without prior anticancer treatment will be treated with antitumor medication. But since BCC is mainly localized in clearly visible regions of the body, as e.g. the face, there is also a need to reduce scars as a consequence of surgery which will be accomplished by neoadjuvant therapy.

The used medication - vismodegib - displays controllable adverse events and shows a good efficacy for reduction of BCC lesions. It is expected that the neoadjuvant setting will lead to minor surgical intervention thus minimising surgical risks and scars for the patients.

DETAILED DESCRIPTION:
Patients with resectable BCC will receive neoadjuvant vismodegib therapy for a time period of 12 weeks which applies to the routine use of vismodegib. This period is chosen because within this time side effects are acceptable and response is expected. Tumor examination will be performed monthly to expeditiously identify patients with progressive disease. This will be done by non-invasive imaging techniques thus a further objective of this study is the testing of diagnostic suitability of non-invasive methodology for the evaluation of response status of the patients.

Patients in this clinical trial will be treated with an effective medication which is approved for the therapy of metastatic and locally advanced BCC for a time having been shown to be effective in neoadjuvant setting The same dose as approved for the advanced BCC disease is used, therefore it can be expected that the side effects will be predictable. Furthermore there are no hints in literature that the efficacy of the used medication may be decreased in patients with resectable BCC.

Since the study patients are less sick than those for whom treatment with vismodegib is approved, surgery would be their therapy according to guideline. Thus the risk of vismodegib treatment has to be judged against the greater surgical risk if BCC will be operated directly without prior reduction of tumor lesion. A benefit for the great majority of the patients will be that smaller lesions result in minor scars and better cosmetically outcome of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged ≥ 18 years
2. Able to participate and willing to give written informed consent including consent for photographs prior to performance of study-related procedures and to comply with the study protocol.
3. Patients with at least 1 large (≥ 2 cm in diameter in head/neck region, ≥ 5 cm for trunk/extremities) basal cell carcinoma (BCC), still resectable, but with increased risk for cosmetic disfigurement or functional defects by assessment of the enrolling physician. Patients with large (as defined above) recurrent basal cell carcinoma are also eligible.
4. Patients must be naïve to treatment with vismodegib or other hedgehog pathway inhibitors
5. Local histopathologic confirmation of BCC (3 mm punch biopsy)
6. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
7. Consent to undergo mapping biopsies upon reaching complete response

   Adequate hematologic and organ function, defined by the following laboratory results, to be obtained within 7 days prior to registration and prior to first dose of study drug treatment:
   * Absolute neutrophilic count > 1,0 x 109/L
   * Platelet count ≥ 75 x 109/L
   * Hemoglobin ≥ 8,5 g/dL
   * Albumin ≥ 2.5 g/dL
   * Bilirubin ≤ 1.5 x the upper limit of normal (ULN) or within 3 x ULN for patients
   * Aspartate-aminotransferase, Alanine-aminotransferase, and alkaline phosphatase ≤ 3 x ULN
   * Serum creatinine ≤ 1.5 x ULN
8. Female patients of childbearing potential must agree to always use 2 effective forms of contraception including one highly effective method and a barrier method during treatment with study medication and for 24 months after the final dose. Male patients with partners of childbearing potential must always use a condom (with spermicide, if available), even after a vasectomy, during treatment with study medication and for at least 2 months after the final dose. Breast feeding is likewise not allowed for at least 24 months after completion of study therapy.
9. Negative serum pregnancy test within 7 days prior to commencement of dosing in women of childbearing potential (including pre-menopausal women with tubal ligation).
10. Absence of any psychological, familial, sociological, or geographical condition that potentially hampers compliance with the study protocol and follow-up as defined by the treatment discontinuation schedule.
11. Agreement not to donate blood or blood products during the study and for at least 24 months after discontinuation of vismodegib. Because vismodegib has been detected in seminal fluid, in addition for men, agreement not donate sperm during the study or for at least 2 months after discontinuation of therapy
12. Optional: Consent to undergo non-invasive imaging examinations by means of confocal laserscan-microscopy (CLSM) and/or optical coherence tomography (OCT), during and after end of study treatment.

Exclusion Criteria:

1. History of prior treatment with vismodegib or any other hedgehog pathway inhibitor.
2. Radiotherapy that involved the field of the target lesion within 6 months prior to registration. Only one radiotherapy of the target lesion performed > 6 months prior to registration is allowed. If a second radiotherapy in this field took place, patient will be excluded.
3. Any metastatic BCC
4. BCC lesion that is considered to be inoperable (e.g. medical contraindication to surgery, suspicion of bone infiltration)
5. Metatypic BCC
6. Known or suspected Gorlin-Goltz syndrome
7. Uncontrolled medical illness, including advanced malignancies (no activities of the malignancies in the past 3 years), at the discretion of the Investigator
8. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect interpretation of the results of the study or renders the patient at high risk for treatment complications
9. History (within 6 months prior to registration) or current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
10. Any medical or psychological illness or condition preventing adequate consent or ability to comply with the protocol
11. Inability or unwillingness to swallow capsules
12. Inability or unwillingness to comply with study and follow-up procedures
13. Current severe, uncontrolled systemic disease
14. History of malabsorption or other conditions that would interfere with the absorption of the orally applicated study drug
15. Pregnant, lactating, or breast feeding women
16. Patients with one of the following rare hereditary conditions: galactose intolerance, primary hypolactasia, or glucose-galactose malabsorption
17. Participation in another clinical study within 28 days before registration or within a time period of five elimination half-lives of the slowest eliminated previously used study drug (whichever is the longest time period).
18. Known or suspected alcohol or drug abuse in the opinion of the investigator
19. Known hypersensitivity reaction to vismodegib or any of the other ingredients of this medicine
20. Treatment with St John's wort (Hypericum perforatum)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01; Primary Completion 2020-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Disease control rate (DCR) defined as complete response (CR), partial response (PR), or stable disease (SD) after 12 weeks of treatment with vismodegib | 12 weeks
  Rate of patients with CR, PR and SD
Objective and relative (%) reduction of the involved skin surface after 12 weeks of treatment with vismodegib | 12 weeks
  Percent change of the BCC area from baseline to end of study therapy

SECONDARY OUTCOMES:
DCR (CR, PR, or SD) after 12 weeks of treatment with vismodegib in the neoadjuvant treatment setting for different basal cell carcinoma histotypes (superficial, scleroderma, nodular, others) | 12 weeks
Duration of overall response (DoR) | 12 months
  Time from documented CR, PR or SD until progression of disease
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 12 months
Health-related quality of life in patients receiving vismodegib for neoadjuvant treatment of basal cell carcinoma as measured by the Skindex-16 questionnaire | 12 months

OTHER OUTCOMES:
Diagnostic suitability of non-invasive imaging techniques (in vivo confocal laserscan-microscopy and/or optical coherence tomography for the evaluation of response status of patients receiving vismodegib in the neoadjuvant setting) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kaatz, PD Dr., Principal Investigator — martin.kaatz@wkg.srh.de
Locations (12):
- Germany (12):
  - SRH Wald-Klinikum Gera GmbH, Gera, Thuringia
  - Klinikum Augsburg Süd, Augsburg
  - Charité - Universitätsmedizin Berlin, Berlin
  - Elbe Kliniken Stade - Buxtehude GmbH, Buxtehude
  - Universitätsklinik Carl Gustav Carus der Technischen Universität Dresden, Dresden
  - HELIOS Klinikum Erfurt, Erfurt
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Münster, Münster
  - Fachklinik Hornheide, Münster
  - Klinikum Nürnberg Nord, Nuremberg
  - Harzklinikum Dorothea Christiane Erxleben GmbH, Quedlinburg
  - Universitätsklinikum Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lauterbach B, Kakkassery V, Debus D, Heindl LM, Schultz ES. [Advanced periocular basal cell carcinoma-a therapeutic challenge]. Ophthalmologe. 2019 Mar;116(3):273-277. doi: 10.1007/s00347-018-0734-9. German. PMID 29777299